CLINICAL TRIAL: NCT03700710
Title: Remote Dietary Counseling Using Web-based Tools to Promote Healthy Diet and Blood Pressure (Healthy BP)
Brief Title: Remote Dietary Counseling to Promote Healthy Diet and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0433
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Blood Pressure; High Blood Pressure; Dietary Modification; Overweight and Obesity
Keywords: lifestyle modification; DASH diet; weight loss; exercise
MeSH Terms: conditions — Hypertension; Overweight; Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Guided Approach (Active Comparator): In the self-guided arm, participants will receive access to web-based tools to help achieve healthy lifestyle changes to lower their blood pressure.
  The web-based tools include: 1) a web-based food frequency questionnaire (Viocare FFQ), which will provide a snapshot of participants' dietary habits in the past 6 months as well as personalized recommendations for areas to improve; 2) access to an evidence-based program (Evolve, formerly BMIQ), which includes program materials for weight loss and leading a healthy lifestyle as well as the ability for capturing dietary data entry.
  Interventions: Behavioral: Self-Guided Approach
- Dietitian-led Approach (Experimental): In the dietitian-led arm, dietitian will use motivational interviewing in 15-30 minute telephone calls with participants.
  The web-based tools include: 1) a web-based food frequency questionnaire (Viocare FFQ), which will provide a snapshot of participants' dietary habits in the past 6 months as well as personalized recommendations for areas to improve; 2) access to an evidence-based program (Evolve, formerly BMIQ), which includes program materials for weight loss and leading a healthy lifestyle as well as the ability for capturing dietary data entry.
  The web platform will be used to share participant dietary and weight data with dietitians.
  Interventions: Behavioral: Dietitian-led Approach

INTERVENTIONS:
Behavioral: Self-Guided Approach — For a 12-week period, patients will be asked to access the web platform (Evolve, formerly BMIQ), review educational materials, and enter dietary information.
  From January 2019 to February 2021, participants used an earlier version of the platform, which was used in tandem with LoseIt (www.loseit.com), a meal-logging app that integrated with the platform.
  In February 2021, a platform update occurred (Evolve) where the core tenets of the program remained the same and included the dietary data entry directly on the platform.
  Arms: Self-Guided Approach
Behavioral: Dietitian-led Approach — For a 12-week period, patients will be asked to access the web platform (Evolve, formerly BMIQ), review educational materials, and enter dietary information.
  From January 2019 to February 2021, participants used an earlier version of the platform, which was used in tandem with LoseIt (www.loseit.com), a meal-logging app that integrated with the platform.
  In February 2021, a platform update occurred (Evolve) where the core tenets of the program remained the same and included the dietary data entry directly on the platform.
  Dietitians will access the web platform and provided personalized motivational interview phone calls on a weekly basis.
  Arms: Dietitian-led Approach

SUMMARY:
American College of Cardiology/American Heart Association (ACC/AHA) hypertension guidelines recommend lifestyle modification for patients with elevated blood pressure. While eating a Dietary Approaches to Stop Hypertension (DASH)-type diet, increasing physical activity, and weight loss have been shown to reduce blood pressure, limited resources are available in the primary care setting to help patients make these changes.

In this study, the investigators will compare the efficacy of a self-guided vs. dietitian-led approach using web-based lifestyle modification tools to reduce weight, improve dietary quality, and lower blood pressure in overweight/obese adults with elevated blood pressure.

DETAILED DESCRIPTION:
Goals that all participants will be instructed to target include: 1) weight loss >=3% at 3 months; 2) consume a healthier dietary pattern (high in fruits, vegetables, whole grains, low-fat dairy, vegetable/fish/poultry sources of protein, healthier sources of fat, and avoid sugar and salt); 3) reduce sodium intake to <2300 mg/d; 4) at least 180 min/wk of moderate-intensity physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 24-hour ambulatory SBP 120-160 mmHg
* BMI ≥ 25 kg/m2
* Access to a telephone
* Access to a computer or smartphone with internet access
* Complete dietary data entry for at least 5 out of 7 days during run-in period
* Enter weight into the platform during run-in period

Exclusion Criteria:

* Inability to understand English
* Myocardial infarction, stroke, or atherosclerotic cardiovascular disease procedure within last 6 months.
* Current treatment for malignancy
* Planned or previous bariatric surgery
* Pregnant, breast-feeding, or planned pregnancy prior to the end of participation
* Self-reported average consumption of > 21 alcoholic beverages per week or binge drinking.
* Psychiatric hospitalization in past year
* Current symptoms of angina
* Planning to leave the area prior to end of the study
* Current participation in another clinical trial
* Principal investigator discretion (i.e. concerns about safety, compliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour Systolic Blood Pressure | Baseline to 12-week follow-up
  Measured by 24-hour ambulatory blood pressure monitoring (SpaceLabs Ontrak)

SECONDARY OUTCOMES:
Change in 24-hour diastolic blood pressure | Baseline to 12-week follow-up
  Measured by 24-hour ambulatory blood pressure monitoring (SpaceLabs Ontrak)
Change in Daytime Systolic Blood Pressure | Baseline to 12-week follow-up
  Measured by 24-hour ambulatory blood pressure monitoring (SpaceLabs Ontrak)
Change in Nighttime Systolic Blood Pressure | Baseline to 12-week follow-up
  Measured by 24-hour ambulatory blood pressure monitoring (SpaceLabs Ontrak)
Change in Daytime Diastolic Blood Pressure | Baseline to 12-week follow-up
  Measured by 24-hour ambulatory blood pressure monitoring (SpaceLabs Ontrak)
Change in Nighttime Diastolic Blood Pressure | Baseline to 12-week follow-up
  Measured by 24-hour ambulatory blood pressure monitoring (SpaceLabs Ontrak)
Change in Total Healthy Eating Index - 2015 score | Baseline to 12-week follow-up
  Assessed by Viocare Food Frequency Questionnaire (score 0-100, 100=best possible score)
Change in Weight | Baseline to 12-week follow-up
  Weight measured at baseline and 12-week visits without shoes
Change in Waist Circumference | Baseline to 12-week follow-up
  Measured using a tape measure
Change in Physical Activity (metabolic equivalent of task [MET]-minute per week | Baseline to 12-week follow-up
  Measured by International Physical Activity Questionnaire (IPAQ) Short Form

OTHER OUTCOMES:
Change in individual components of Healthy Eating Index score | Baseline to 12-week follow-up
  Each individual component of the Healthy Eating Index score will be examined
Satisfaction with the Healthy BP Research Study | 12-week follow-up
  5-point Likert score

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chang, MD, Principal Investigator — Geisinger Clinic
Locations (2):
- United States (2):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, informed consent form, analytic code, and clinical study report will be shared at the time of publication of the main trial results; these data will be deidentified. These data will be publicly available indefinitely.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the time of publication of the main trial results and will be publicly available indefinitely.
Access Criteria: The deidentified IPD will be publicly available without restrictions.

REFERENCES:
- [Derived] Chang AR, Gummo L, Yule C, Bonaparte H, Collins C, Naylor A, Appel LJ, Juraschek SP, Bailey-Davis L. Effects of a Dietitian-Led, Telehealth Lifestyle Intervention on Blood Pressure: Results of a Randomized, Controlled Trial. J Am Heart Assoc. 2022 Oct 4;11(19):e027213. doi: 10.1161/JAHA.122.027213. Epub 2022 Sep 29. PMID 36172955
- [Derived] Taher M, Yule C, Bonaparte H, Kwiecien S, Collins C, Naylor A, Juraschek SP, Bailey-Davis L, Chang AR. Telehealth versus self-directed lifestyle intervention to promote healthy blood pressure: a protocol for a randomised controlled trial. BMJ Open. 2021 Mar 3;11(3):e044292. doi: 10.1136/bmjopen-2020-044292. PMID 33658261